CLINICAL TRIAL: NCT07227220
Title: Leveraging Summer Youth Employment Programs to Prevent Obesity in Adolescents
Brief Title: Summer Youth Employment Programs for Health Promotion
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Houston (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00005180
Record Dates: First submitted 2025-08-04; First posted 2025-11-12 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-10

CONDITIONS: Obesity, Childhood; Behavior, Health; Healthy Lifestyle
MeSH Terms: conditions — Pediatric Obesity; Health Behavior

STUDY DESIGN:
Intervention Model Description: Single group pre- and post-test design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Summer Youth Employment Program (Experimental): Participants will work as junior summer camp counselors at a University of Houston camp, up to 24 hours/week, Monday-Thursday, 8:30 AM-3:30 PM (with a 12-1 PM lunch break), for six weeks from mid-June to the end of July. Participants will assist senior counselors with indoor/outdoor activities such as games, enrichment, and academics. On Fridays, from 10 AM to 12 PM, participants will attend professional development workshops on topics such as communication, teamwork, resume building, and job search skills. From 12-2:30 PM, undergraduate staff will lead social activities and mentoring.
  Interventions: Behavioral: Summer Youth Employment Program

INTERVENTIONS:
Behavioral: Summer Youth Employment Program — The intervention aims to employ adolescents in paid positions for six weeks during the summer, providing them with a structured, routine-based, and adult-supervised environment similar to that of the school year.

SUMMARY:
The purpose of this proof-of-concept study is to assess the initial signal of effectiveness of summer youth employment programs (SYEP) on understudied obesity-related outcomes in adolescents. This small-scale study is essential to identify early success and refine the intervention before scaling to a larger, more resource-intensive randomized trial. Specifically, this one-group pre-posttest study will:

Aim 1 (Primary): Evaluate if a 6-week SYEP provides an initial signal for effectiveness (maintenance or decrease in zBMI) over the summer.

Hypothesis 1: Adolescents who participated in a SYEP will maintain or decrease their BMI over the summer.

Aim 2 (Secondary): Evaluate changes in obesogenic behaviors (physical activity, sleep, sedentary, and diet) over the summer.

Hypothesis 2: Adolescents who participated in a SYEP will increase physical activity, reduce sedentary behavior, and improve sleep and diet quality over the summer.

Aim 3 (Secondary): Evaluate the feasibility of SYEP for obesity prevention intervention to inform intervention scalability.

Hypothesis 3: The SYEP program will be a feasible and acceptable intervention strategy for the prevention of obesity in adolescents over the summer.

DETAILED DESCRIPTION:
Preliminary evidence suggests that summer employment can be an age-appropriate, structured intervention to prevent unhealthy changes in obesogenic behaviors among adolescents. While these findings are promising, none of the existing studies have measured changes in BMI over the summer or conducted comprehensive assessments of obesogenic behaviors, including diet, sedentary behavior, sleep, and physical activity. To address these gaps, this study proposes a small proof-of-concept study to assess the initial signal of effectiveness on understudied obesity-related outcomes in adolescents.

SYEPs are well-established, continuously operating initiatives over 60 years with proven benefits in academics, workforce development, and crime prevention, and may also act as obesity prevention strategies. Rather than creating new interventions, investing in and expanding access to SYEPs-programs with high demand yet limited capacity (with only ~28% of applicants matched with jobs each summer, leaving the majority on waitlists)-can offer a practical solution for youth obesity prevention.

ELIGIBILITY:
Inclusion Criteria:

* Age 14-17 years at the time of enrollment, in accordance with Texas Child Labor Law
* Willing to work at the summer camp for six consecutive weeks
* Able to pass the employment admission procedure (job interview)
* Able to obtain parental consent and provide assent for study participation

Exclusion Criteria:

* Currently pregnant or planning to become pregnant, due to physical activity restrictions and potential weight changes that could confound study results
* Diagnosis of an intellectual and/or physical disability requiring specialized employment regulations or intervention strategies
* Participation in a health promotion intervention within the past six months

Ages: 14 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 2025-03-31 (Actual); Primary Completion 2025-07-07 (Actual); Study Completion 2025-07-29 (Actual)

PRIMARY OUTCOMES:
zBMI | Baseline and Week 6 (post)
  Height and weight will be directly measured by trained staff. Each measurement will be taken twice, and the average will be used for analysis. Changes in BMI will be expressed as Centers for Disease Control age-sex specific z-scores (zBMI).

SECONDARY OUTCOMES:
Sedentary behaviors | Baseline and Week 6 (post)
  Sedentary behavior (minutes per day) will be measured using a wrist-placed ActiGraph GT3X on the non-dominant wrist for 8 days, ensuring at least 2 valid weekdays and 1 weekend. Cut points published by Hildebrand et al. will be used to classify activity intensities.
Moderate to vigorous physical activity (MVPA) | Baseline and Week 6 (post)
  MVPA (minutes per day) will be measured using a wrist-placed ActiGraph GT3X on the non-dominant wrist for 8 days, ensuring at least 2 valid weekdays and 1 weekend. Cut points published by Hildebrand et al. will be used to classify activity intensities.
Sleep Duration | Baseline and Week 6 (post)
  Sleep duration (minutes per day) will be measured using a wrist-placed ActiGraph GT3X on the non-dominant wrist for 8 days, ensuring at least 2 valid weekdays and 1 weekend. Sleep duration will be determined using the heuristic algorithm looking at distribution of change in Z-Angle (HDCZA).
Screen Time | Baseline and Week 6 (post)
  Screen time in hours and minutes (e.g., television, computer, video games, smart phones, tablets) will assessed via self-report during each 8-day behavioral assessment period. Daily average screen time duration in minutes will be calculated by summing the total screen time across completed daily logbooks and dividing by the number of days the diary was completed.
Diet Intake | Baseline and Week 6 (post)
  Adolescents will self-report their dietary intake via NHANES 23-item Dietary Screener Questionnaire. Responses will be dichotomized based on their distribution into two categories: "did not eat/drink today" and "ate/drank today". Subsequently, items will be grouped into two broader categories: healthy foods (fruits, vegetables, 100% fruit juice, and milk items) and unhealthy foods (desserts, sugar-sweetened beverages, salty snacks, and fast food items).
Recruitment capacity (percentage meeting recruitment goal) | Baseline
  Recruitment capacity is the percentage meeting the recruitment goal.
Retention | Baseline and Week 6 (post)
  Retention (primary outcome) is the proportion of enrolled participants who completed both baseline and post-assessments for the primary outcome.
Fidelity | Weekly during intervention (Weeks 1-6)
  Investigators will measure fidelity through weekly direct observations using a short checklist to record content delivery with time logs and supervisor behaviors.
Attendance | Weekly during intervention (Weeks 1-6)
  Attendance will be tracked as the proportion of days attended out of total offered workdays using employer time sheets.
Acceptability | Week 7 (Follow-up)
  Acceptability will be assessed through individual interviews conducted via Microsoft Teams with adolescents about barriers and facilitators to participation.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Houston, Houston, Texas, United States

REFERENCES:
- [Background] Czajkowski SM, Powell LH, Adler N, Naar-King S, Reynolds KD, Hunter CM, Laraia B, Olster DH, Perna FM, Peterson JC, Epel E, Boyington JE, Charlson ME. From ideas to efficacy: The ORBIT model for developing behavioral treatments for chronic diseases. Health Psychol. 2015 Oct;34(10):971-82. doi: 10.1037/hea0000161. Epub 2015 Feb 2. PMID 25642841
- [Background] Pierce B, Bowden B, McCullagh M, Diehl A, Chissell Z, Rodriguez R, Berman BM, D Adamo CR. A Summer Health Program for African-American High School Students in Baltimore, Maryland: Community Partnership for Integrative Health. Explore (NY). 2017 May-Jun;13(3):186-197. doi: 10.1016/j.explore.2017.02.002. Epub 2017 Feb 24. PMID 28373062
- [Background] Yazel-Smith L, El-Mikati HK, Adjei M, Haberlin-Pittz KM, Agnew M, Hannon TS. Integrating Diabetes Prevention Education Among Teenagers Involved in Summer Employment: Encouraging Environments for Health in Adolescence (ENHANCE). J Community Health. 2020 Aug;45(4):856-861. doi: 10.1007/s10900-020-00802-2. PMID 32146639
- [Background] Modestino AS, Paulsen RJ. Reducing inequality summer by summer: Lessons from an evaluation of the Boston Summer Youth Employment Program. Eval Program Plann. 2019 Feb;72:40-53. doi: 10.1016/j.evalprogplan.2018.09.006. Epub 2018 Sep 24. PMID 30296721